CLINICAL TRIAL: NCT05534529
Title: A Phase 1, Multicentre, Open-Label Study to Evaluate the PK, Safety, and Tolerability of a Single IV Dose of Rezafungin in Paediatric Subjects, Receiving Systemic Antifungals as Prophylaxis for IFI or to Treat a Suspected or Confirmed FI
Brief Title: Rezafungin Paediatric PK Study in Paediatric Subjects From Birth to <18 Years of Age
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The study had initially anticipated dosing of the first cohort within 4-9 months of activation; however the study faced significant challenges in recruitment. In order to adhere to the previously approved PIP plan, the study could not be redesigned.
Sponsor: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MR907-1501
Record Dates: First submitted 2022-09-01; First posted 2022-09-09 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Invasive Fungal Infections
Keywords: Rezafungin, children and adolescents, systemic anti-fungal treatment; Pharmacokinetics
MeSH Terms: conditions — Invasive Fungal Infections | interventions — Rezafungin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Rezafungin (Experimental): It is IMP.
  Interventions: Drug: Rezafungin Acetate

INTERVENTIONS:
Drug: Rezafungin Acetate — This is a Phase 1, multicentre, open-label, single-dose study. The study will be conducted at 10 sites across at least 3 countries in Europe.
  Other Names: Rezafungin

SUMMARY:
This study aimed to learn what levels of rezafungin were in the blood after dosing and how safe it was, in children and adolescents below 18 years old who were already receiving treatment for a fungal infection, a suspected fungal infection or at risk of fungal infection.

The main question the researchers wanted to answer in this trial was:

• What were the levels of rezafungin in the blood after the participants were dosed? The researchers also wanted to know what medical problems happened during this trial.

The participants in this trial received one dose of rezafungin on day 1 through a needle into a vein, called an intravenous (IV) infusion. The dose of rezafungin was measured in milligrams (mg) and given to the participants according to their body weight in kilograms (mg/kg).

The doctors checked the participants' health and asked questions about what medications they were taking and took blood samples to check the levels of rezafungin in the participants' blood.

After receiving the treatment at day 30, the doctors checked the participants' health.

This was an "open-label" trial. This means each participant knew what they were receiving, and the doctors and trial staff also knew.

DETAILED DESCRIPTION:
To date, there are no clinical studies evaluating rezafungin in paediatric subjects.

The primary objective of the trial was to evaluate the pharmacokinetics (PK) of a single intravenous (IV) dose of rezafungin in paediatric participants from birth to < 18 years, receiving concomitant systemic antifungals as prophylaxis for invasive fungal infection (IFI) or to treat a suspected or confirmed fungal infection.

The secondary objective was to assess the safety and tolerability of a single IV dose of rezafungin in the subjects.

This is a Phase 1, multicentre, open-label, single-dose study. The study will be conducted at approximately 10 sites across at least 3 countries in Europe.

The study will be conducted in 3 parts:

* Part 1 will include subjects aged 12 to <18 years (Group 1)
* Part 2 will include subjects aged 6 to <12 years (Group 2), and subjects aged 2 to <6 years (Group 3).
* Part 3 will include subjects from birth to <2 years (Group 4) The study design for the 3 parts is similar and comprises a Screening (pre-treatment) period from Day -3 to Day -1, Dosing on Day 1 (single IV infusion of rezafungin) followed by multiple PK sampling, and a Follow up visit on Day 30 (± 5 days). PK sampling will be performed at specified timepoints for each group.

Limitations and Caveats Due to recruitment challenges, the study was terminated following enrollment of 2 participants aged between 12-17 years in Group 1 (Part 1). Group 2, 3 (Part 2) and Group 4 (Part 3) were not initiated prior to study termination. Due to the low number of participants in this study, baseline characteristics, outcome measure results and adverse events have not been reported to reduce the potential of re-identification.

ELIGIBILITY:
Inclusion Criteria:

* Male or female paediatric subjects from birth to <18 years of age who are receiving concomitant systemic antifungals (oral or IV) as prophylaxis for invasive fungal infection (IFI) or to treat a suspected or confirmed fungal infection.

Exclusion Criteria:

* History of anaphylaxis, hypersensitivity, or any serious reaction to the echinocandin class of antifungals and/or excipients of this formulation
* Previous or current medical conditions of severe ataxia, persistent tremors, intracranial hemorrhage or neuropathy, or a diagnosis of epilepsy, multiple sclerosis, or a movement disorder
* Subjects with impaired renal or hepatic functions
* Subjects with intestinal hypoxia, ischemia, necrosis, or necrotizing enterocolitis
* Subject status is unstable
* Subject is unlikely to complete required study procedures
* Participation in another interventional treatment trial with an investigational agent or presence of an investigational device at the time of informed consent or within 28 days preceding the informed consent.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 32 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Rezafungin | At end-of-infusion ± 15 minutes, then between 3 and 4 hours after start of infusion, between 6 and 8 hours after start of infusion, at 48 hours (± 4 hours) after start of infusion, and at 168 hours (± 12 hours) after start of infusion
  Blood samples of 1 mL each were collected for the analysis of rezafungin plasma concentration. PK parameters were determined from the rezafungin concentration-time data using non-compartmental methods and actual sampling times.
Time at which the Cmax of Rezafungin Was Observed (Tmax) | End of infusion and 3-4, 6-8, 48, and 168 hours after start of infusion
  Blood samples of 1 mL each were collected for the analysis of rezafungin plasma concentration. PK parameters were determined from the rezafungin concentration-time data using non-compartmental methods and actual sampling times.
Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration (AUC0-t) of Rezafungin | End of infusion and 3-4, 6-8, 48, and 168 hours after start of infusion
  Blood samples of 1 mL each were collected for the analysis of rezafungin plasma concentration. PK parameters were determined from the rezafungin concentration-time data using non-compartmental methods and actual sampling times.
Area Under the Plasma Concentration-time Curve From Time 0 Extrapolated to Infinity (AUC0-∞) of Rezafungin | End of infusion and 3-4, 6-8, 48, and 168 hours after start of infusion
  Blood samples of 1 mL each were collected for the analysis of rezafungin plasma concentration. PK parameters were determined from the rezafungin concentration-time data using non-compartmental methods and actual sampling times.
Total Clearance (CL) of Rezafungin | End of infusion and 3-4, 6-8, 48, and 168 hours after start of infusion
  Blood samples of 1 mL each were collected for the analysis of rezafungin plasma concentration. PK parameters were determined from the rezafungin concentration-time data using non-compartmental methods and actual sampling times.
Volume of Distribution of Rezafungin at Steady-state (Vss) | End of infusion and 3-4, 6-8, 48, and 168 hours after start of infusion
  Blood samples of 1 mL each were collected for the analysis of rezafungin plasma concentration. PK parameters were determined from the rezafungin concentration-time data using non-compartmental methods and actual sampling times.
Apparent Volume of Distribution of Rezafungin During the Terminal Phase (Vz) | End of infusion and 3-4, 6-8, 48, and 168 hours after start of infusion
  Blood samples of 1 mL each were collected for the analysis of rezafungin plasma concentration. PK parameters were determined from the rezafungin concentration-time data using non-compartmental methods and actual sampling times.
Terminal Elimination Half-life of Rezafungin (t1/2) | End of infusion and 3-4, 6-8, 48, and 168 hours after start of infusion
  Blood samples of 1 mL each were collected for the analysis of rezafungin plasma concentration. PK parameters were determined from the rezafungin concentration-time data using non-compartmental methods and actual sampling times.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | From start of study on Day 1 to follow up Day 30 (+/- days)
  A TEAE was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of rezafungin, whether or not considered related to the rezafungin that was not present prior to the administration of rezafungin or any event present that worsened in either severity or frequency following exposure to rezafungin.
  Clinically significant changes in laboratory evaluations (including haematology, blood chemistry and urinalysis), vital signs, 12-lead electrocardiogram (ECG) and physical examination findings were also reported as TEAEs.

CONTACTS AND LOCATIONS:
Locations (10):
- Germany (3):
  - Universitätsklinikum Essen Zentrum für Kinder- und Jugendmedizin, Essen
  - Universitätsklinikum Frankfurt, Goethe Universität Klinik für Kinder- und Jugendmedizin, Frankfurt
  - Universitätsklinikum Münster Klinik für Kinder- und Jugendmedizin, Münster
- Spain (3):
  - Hospital Universitario de Burgos, Burgos
  - Hospital Universitario 12 de Octubre., Madrid
  - Hospital Universitario La Paz, Madrid
- United Kingdom (4):
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - Saint Mary's Hospital, Imperial College Healthcare NHS Trust, London
  - St. George's University Hospitals, NHS Foundation Trust, London
  - Southampton General Hospital, University Hospital Southampton NHS Foundation Trust, Southampton

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-18): https://cdn.clinicaltrials.gov/large-docs/29/NCT05534529/Prot_SAP_000.pdf